CLINICAL TRIAL: NCT07036393
Title: Acupuncture Versus Transcutaneous Electrical Nerve Stimulation on Pain Post Upper Abdominal Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Saad Nazim Mohamed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Samar-005748
Record Dates: First submitted 2025-06-14; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acupuncture; Transcutaneous Electrical Nerve Stimulation; Pain; Upper Abdominal Surgery
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy; Transcutaneous Electric Nerve Stimulation; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): This group includes 20 patients who will receive Acupuncture 4 weeks (3times/week) and medical treatment
  Interventions: Other: Acupuncture; Other: drugs
- Transcutaneous electrical nerve stimulation (Active Comparator): This group includes 20 patients who will receive Transcutaneous electrical nerve stimulation 4 weeks (3times/week) and medical treatment
  Interventions: Other: Transcutaneous electrical nerve stimulation; Other: drugs

INTERVENTIONS:
Other: Acupuncture — Cholecystectomy involves a procedure where patients' spines are kept in position and skin around the acupoints is disinfected with 75% alcohol. Acupuncture treatment is given when patients return to units within 2 hours after surgery. The needles are inserted using disposable sterile needles and manipulated to induce a sense of "De qi" (soreness, numbness, distension, or heaviness). Gastrectomy involves daily acupuncture sessions for 5 consecutive days, starting on postoperative day 1. The needles are inserted perpendicular to the acupoints in the extremities to a depth of approximately 20 mm from the skin surface.
  Arms: Acupuncture
Other: Transcutaneous electrical nerve stimulation — Patients will receive a transcutaneous electrical nerve stimulation unit (ENNRAF) for up to 48 hours post-surgery, with instructions to self-titrate intensity for pain relief. Postoperative stimulation will be 20-40 milliampere and pulse width 5
  Arms: Transcutaneous electrical nerve stimulation
Other: drugs — analgesics and nonsteroidal anti-inflammatory drugs

SUMMARY:
This study was done to:

* Determine the therapeutic efficacy of acupuncture as physical therapy approach in minimizing pain post upper abdominal surgeries.
* Determine the therapeutic efficacy of transcutaneous electrical nerve stimulation in minimizing pain post upper abdominal surgeries.
* Compare the efficacy and safety of Transcutaneous electrical nerve stimulation versus acupuncture in minimizing pain post upper abdominal surgeries.

DETAILED DESCRIPTION:
Postoperative pain is caused by tissue damage from surgical incisions, triggering acute nociceptive activity in sensory nerve endings. Pain sensations reach the brain through dorsal horn, where it is recognized and interpreted. Management modalities include pharmacologic and non-pharmacologic methods. This study aims to provide a guideline on the effect of acupuncture and transcutaneous electrical nerve stimulation on pain reduction after upper abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will have pain after upper abdominal surgery.
* Adult patients will be between 20 and 45 years of age.
* Both sexes will be included.
* Patients have no contraindications for acupuncture or transcutaneous electrical nerve stimulation.
* Patients with good compliance and fit for treatment.
* This study will be applied on upper abdominal surgeries [laparoscopic cholecystectomy, Gastrectomy].
* Physical therapy will be used for up to 48 hours after surgery or until the time of discharge.

Exclusion Criteria:

* Patients with other causes of pain other than that after upper abdominal surgery.
* Patients who will have any contraindication for both therapies used.
* Patients with cardiovascular disease, liver, or renal disease.
* Patients with malignant tumors.
* Patients with metal or electronic implants.
* Patients with autoimmune disease.
* Pregnancy, postpartum period, breastfeeding.
* Patients with recent injury in the treatment area

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
assessment of change of postoperative quality of recovery | At baseline and 4 weeks
  The Postoperative Quality of Recovery Scale is a verbal scale designed to assess the quality of recovery in six domains: physiology, nociceptive, emotional, activities of daily living, cognitive, and overall patient perspective. It measures systolic blood pressure, heart rate, temperature, respiratory rate, oxygen saturation, and airway control, aiming to assess physiologic safety and home readiness for day care surgery. It also assesses pain and nausea using a 1-5% Likert rating scale. Emotional domain measures feelings of anxiety and depression. Activities of daily living assess physical return to normality through daily activities, with scores ranging from 3 to 1. Cognitive domain measures orientation, verbal memory, executive functioning, attention, and concentration. Performance variability tolerance factors are applied to ensure participants are not included in subsequent analysis if baseline scores are equal to or less than the tolerance factor.

SECONDARY OUTCOMES:
assessment of change of pressure pain threshold | At baseline and 4 weeks
  An algometer is a handheld device used for pressure tolerance testing, typically with a 1-cm2 pressure application surface and force readings in newtons or kilograms. It has a resolution of 0.2 newton, 250-newton capacity, and a 1000-Hz sampling rate. The device is designed to measure pains and track recovery/healing, and is tested for high reliability and validity compared to force plate readings.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura international hospital, Al Mansurah, Egypt